CLINICAL TRIAL: NCT02038647
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Clinical Trial of Alisertib (MLN8237) in Combination With Paclitaxel Versus Placebo in Combination With Paclitaxel as Second Line Therapy for Small Cell Lung Cancer (SCLC).
Brief Title: Phase 2 Study of Alisertib (MLN8237) in Combination With Paclitaxel Versus Placebo in Combination With Paclitaxel as Second Line Therapy for Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C14018; 2013-003713-18 (EudraCT Number); U1111-1154-9805 (Registry Identifier: WHO); DRKS00007849 (Registry Identifier: DRKS)
Record Dates: First submitted 2013-12-04; First posted 2014-01-16 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Drug therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — MLN 8237; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alisertib (MLN8237) + Paclitaxel (Experimental): Alisertib 40 mg, tablets, orally, twice a day, 3 days on/4 days off for 3 weeks on Days 1-3, 8-10, and 15-17 in a 28-day cycle along with paclitaxel 60 mg/m^2 intravenously (IV) once a week for 3 weeks on Days 1, 8, and 15 in a 28-day until disease progression (Up to 17 Cycles).
  Interventions: Drug: Alisertib; Drug: Paclitaxel
- Placebo + Paclitaxel (Placebo Comparator): Alisertib placebo-matching tablets, orally, twice a day, 3 days on/4 days off for 3 weeks on Days 1-3, 8-10, and 15-17 in a 28-day cycle along with paclitaxel 80 mg/m^2 IV once a week for 3 weeks on Days 1, 8, and 15 in a 28-day cycle until disease progression (Up to 22 Cycles).
  Interventions: Drug: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Drug: Alisertib — Alisertib tablets
  Other Names: MLN8237
  Arms: Alisertib (MLN8237) + Paclitaxel
Drug: Placebo — Placebo matching tablets
  Arms: Placebo + Paclitaxel
Drug: Paclitaxel — Paclitaxel intravenous injection

SUMMARY:
This is a two-arm, randomized, double-blind, placebo-controlled, multicenter, phase 2 study designed to is to determine if the combination treatment can improve progression free survival (defined as the time from the date of randomization to the date of first documentation of disease progression or death, whichever occurs first) when compared with placebo + paclitaxel.

DETAILED DESCRIPTION:
The drug tested in this study is called alisertib. Alisertib is being tested to treat people who have Small Cell Lung Cancer (SCLC). This study determined the safety and efficacy for alisertib when given twice a day along with paclitaxel.

This open label study enrolled 178 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there is an urgent medical need) and participants were stratified at baseline as to whether brain mets were present or not; whether they were sensitive to prior therapy or were relapsed/refractory to prior therapy; and by world region:

* Alisertib 40 mg + Paclitaxel 60 mg/m^2
* Paclitaxel 80 mg/m^2 + Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

All participants received treatment until their disease progressed or they experienced unacceptable alisertib-related toxicity.

This multi-center trial was conducted world-wide. The overall time to participate in this study was approximately up to 22 months. Participants made multiple visits to the clinic, and were contacted by telephone every month for 6 months after the end of treatment (EOT) for follow-up assessment of progression free survival and for overall survival every 2 months until death, study closure, or 14 months after randomization of the last participant.

ELIGIBILITY:
Inclusion Criteria

Each participant must meet all the following inclusion criteria to be enrolled in the study:

1. Male or female participants ≥ 18 years old.
2. Have a pathologically (histology or cytology) confirmed diagnosis of SCLC.
3. Have received and progressed after a platinum-based standard chemotherapy regimen for first line treatment of SCLC, either limited stage (LS) or extensive stage (ES).
4. Have measurable disease within ≤ 2 weeks before randomization. Clear radiographic evidence of disease progression after initial therapy should have been documented.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 (PS 0-1).
6. Participants with treated brain metastases (surgery, whole or stereotactic brain radiation) are allowed provided the lesions have been stable for at least 2 weeks and the participant is off steroids or is on a stable dose of steroids. Participants should be without neurologic dysfunction that would confound the evaluation of neurological and/or other AEs.

Exclusion Criteria

Participants meeting any of the following exclusion criteria are not to be randomized to treatment:

1. Any prior therapy for second-line treatment of SCLC.
2. Participants who relapsed ≥ 180 days after their response to first-line treatment.
3. Prior treatment with an Aurora A specific-targeted or pan-Aurora-targeted agent, including alisertib, or any other investigational agent.
4. Prior treatment with paclitaxel or any other taxane agent.
5. Known hypersensitivity to Cremophor® EL, paclitaxel, or its components.
6. Any comorbid condition or unresolved toxicity that would preclude administration of alisertib or weekly paclitaxel.
7. Prior history of ≥ Grade 2 neurotoxicity that is not resolved to ≤ Grade 1.
8. Participants with symptomatic and/or progressive brain metastases or with carcinomatous meningitis.
9. Treatment with clinically significant enzyme inducers within 14 days prior to the first dose of alisertib and during study conduct. Major prohibited enzyme inducers include: phenytoin, carbamazepine, phenobarbital, rifampin, rifabutin, rifapentine, and St. John's wort.
10. Inability to swallow alisertib or other orally administered medications.
11. Requirement for administration of proton pump inhibitor (PPI), H2 antagonist, or pancreatic enzymes.
12. Diagnosed with or treated for another malignancy within 2 years before the first dose of study drug, or previously diagnosed with another malignancy and have any evidence of residual disease.
13. Other severe acute or chronic medical or psychiatric condition(s) per protocol.
14. History of myocardial infarction, unstable symptomatic ischemic heart disease, uncontrolled hypertension despite appropriate medical therapy, any ongoing cardiac arrhythmias of Grade > 2, thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, or symptomatic cerebrovascular events), or any other cardiac condition (eg, pericardial effusion or restrictive cardiomyopathy) within 6 months before receiving the first dose of study drug.
15. Known history of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C.
16. Surgery within 3 weeks (or 2 weeks for a minor surgery) before study enrollment and not fully recovered to baseline or to a stable clinical status.
17. Participants who are pregnant, lactating, or do not agree to use effective methods of contraception during the study treatment period through 6 months after the last dose of study drug per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2016-01-03 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (61):
- United States (21):
  - Los Angeles, California
  - Sacramento, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Boca Raton, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington
- Belgium (6):
  - Edegem
  - Ghent
  - Kortrijk
  - Leuven
  - Mons
  - Roeselare
- Canada (3):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Greenfield Park
- Czechia (4):
  - Olomouc
  - Ostrava
  - Prague
  - Ústí nad Labem
- France (6):
  - Grenoble
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Rennes
- Germany (4):
  - Berlin
  - Frankfurt
  - Freiburg im Breisgau
  - Lübeck
- Hungary (5):
  - Budapest
  - Farkasgyepű
  - Szolnok
  - Tatabánya
  - Törökbálint
- Italy (3):
  - Milan
  - Orbassano
  - Parma
- Poland (4):
  - Gdansk
  - Mrozy
  - Warsaw
  - Wodzisław Śląski
- Spain (5):
  - A Coruña
  - Barcelona
  - Girona
  - Madrid
  - Seville

REFERENCES:
- [Derived] Owonikoko TK, Niu H, Nackaerts K, Csoszi T, Ostoros G, Mark Z, Baik C, Joy AA, Chouaid C, Jaime JC, Kolek V, Majem M, Roubec J, Santos ES, Chiang AC, Speranza G, Belani CP, Chiappori A, Patel MR, Czebe K, Byers L, Bahamon B, Li C, Sheldon-Waniga E, Kong EF, Williams M, Badola S, Shin H, Bedford L, Ecsedy JA, Bryant M, Jones S, Simmons J, Leonard EJ, Ullmann CD, Spigel DR; C14018 study investigators. Randomized Phase II Study of Paclitaxel plus Alisertib versus Paclitaxel plus Placebo as Second-Line Therapy for SCLC: Primary and Correlative Biomarker Analyses. J Thorac Oncol. 2020 Feb;15(2):274-287. doi: 10.1016/j.jtho.2019.10.013. Epub 2019 Oct 23. PMID 31655296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 54 investigative sites in the United States, Canada, European Union (Belgium, Czech Republic, France, Germany, Hungary, Italy, Poland and Spain) from 12 May 2014 to 10 July 2017. Data cutoff for the primary analysis was 3 January 2016.
Pre-assignment Details: Participants with a diagnosis of Small Cell Lung Cancer (SCLC) were enrolled in 1 of 2 treatment groups: alisertib + paclitaxel or placebo + paclitaxel arm group.
Groups:
- Alisertib + Paclitaxel: Alisertib 40 mg, tablets, orally, twice a day, 3 days on/4 days off for 3 weeks on Days 1-3, 8-10, and 15-17 in a 28-day cycle along with paclitaxel 60 mg/m^2 intravenously (IV) once a week for 3 weeks on Days 1, 8, and 15 in a 28-day cycle until disease progression (Up to 17 Cycles).
Period: Overall Study
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Started | 89 | 89
Completed | 0 | 0
Not Completed | 89 | 89
Not completed — Progressive Disease | 50 | 59
Not completed — Adverse Event | 18 | 10
Not completed — Symptomatic Deterioration | 7 | 7
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Not Reported | 0 | 1
Not completed — Ongoing at Datacut | 9 | 10

BASELINE CHARACTERISTICS:
Population: The ITT population was defined as all participants who were randomized to study treatment, whether or not any treatment was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel | Total
Number analyzed (Participants) | 89 | 89 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (8.55) | 63.4 (8.56) | 62.6 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 51 | 50 | 101
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 81 | 84 | 165
  Unknown or Not Reported | 6 | 1 | 7
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 83 | 83 | 166
  Black or African American | 3 | 2 | 5
  Not reported | 2 | 2 | 4
  Asian | 1 | 0 | 1
  Other | 0 | 1 | 1
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Belgium | 8 | 8 | 16
  Czech Republic | 6 | 5 | 11
  France | 7 | 5 | 12
  Germany | 2 | 1 | 3
  Hungary | 16 | 15 | 31
  Italy | 2 | 0 | 2
  Poland | 1 | 3 | 4
  Spain | 6 | 11 | 17
  Canada | 6 | 6 | 12
  United States | 35 | 35 | 70
Height [Mean (Standard Deviation); unit: cm] — Population: Height data is available for n=86,87 participants respectively.
  cm
    number analyzed (Participants) | 86 | 87 | 173
    (all) | 169.5 (10.43) | 168.8 (9.52) | 169.2 (9.96)
Weight [Mean (Standard Deviation); unit: kg] | 78.47 (20.561) | 75.26 (17.602) | 76.87 (19.153)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area=square root of (height [cm]*weight [kg]/3600). Population: Body Surface Area data is available for n=86,87 participants respectively.
  m^2
    number analyzed (Participants) | 86 | 87 | 173
    (all) | 1.911 (0.2829) | 1.872 (0.2433) | 1.891 (0.2637)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Determined by Investigator, Analyzed Using FDA Guidelines
Description: PFS is defined as time in days from start of study treatment to first documentation of objective tumor progression based on Investigator's assessment or up to death due to any cause, whichever occurs first based on Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. Progressive disease (PD) was defined as ≥20% increase in sum longest diameter (LD) in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Every cycle for first 6 months and then every 2 months until disease progression or death or up to data cut-off: 03 January 2016 (approximately 22 months)
Population: The intent-to-treat (ITT) population was defined as all participants who were randomized to study treatment. For participants who have not progressed and is last known to be alive, PFS was censored at the last response assessment that is stable disease (SD) or better as determined by Investigator, and analyzed using FDA Guidelines.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
days | 101 [80 to 113] | 66 [53 to 83]
Statistical Analysis 1: Comparison: Alisertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.113, Log Rank — P-value tests the hypothesis of equal event times in both treatment arms obtained using the Log-rank test stratified by disease subtype as sensitive versus resistant/refractory and the presence of brain metastases; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.557 to 1.067] — The stratification factors were: disease subtype as sensitive versus resistant/refractory and the presence of brain metastases (yes or no) with treatment (Alisertib + Paclitaxel vs Placebo + Paclitaxel) as a factor in the model

2. Secondary Outcome: Percentage of Participants Who Experience at Least One Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with treatment. An AE can be any unfavorable and unintended sign (eg, clinically significant abnormal laboratory finding), symptom, or disease temporally associated with use of drug, whether or not it is considered related to drug. A treatment-emergent adverse event (TEAE) is defined as an AE with an onset that occurs after receiving study drug. A Serious Adverse Event (SAE) is any experience that suggests significant hazard, contraindication, side effect or precaution that:results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is congenital anomaly/birth defect or is medically significant per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03.
Time Frame: From the first dose through 30 days after the last dose of study medication: data cut-off 03 January 2016 (Up to 10.8 months)
Population: The safety population was defined as all participants who received at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 87 | 89
percentage of participants
  TEAEs | 99 | 96
  SAEs | 44 | 31

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time in days from the date of randomization to the date of death due to any cause.
Time Frame: Contact every 2 months after EOT/disease progression until the sooner of death, study closure, or 14 months after the last participant was randomized up to data cut-off: 3 January 2016 (approximately 22 months)
Population: The ITT population was defined as all participants who were randomized to study treatment. Participants without documentation of death at the time of the analysis were censored at the date when they were last known to be alive.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
days | 186 [150 to 219] | 165 [128 to 183]
Statistical Analysis 1: Comparison: Alisertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.714, Log Rank — [p-value comment as in outcome 1, analysis 1]; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.652 to 1.341] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who achieved CR or partial response (PR) as best response based on Investigator's assessment according to RECIST v 1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as ≥ 30% decrease in sum of LD of target lesions in reference to Baseline sum LD.
Time Frame: Baseline until disease progression, death or EOT up to data cut-off: 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
percentage of participants | 22 [14 to 33] | 18 [11 to 28]
Statistical Analysis 1: Comparison: Alisertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.406, Weighted Cochran-Mantel-Haenszel test — Stratification factors were disease subtypes (sensitive versus resistant/refractory), the presence of brain metastases and region; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.35 to 1.55] — Logistic regression using ORR as dependent variable, treatment arm as independent variable and disease subtype (sensitive vs resistant/refractory) and presence of brain metastases as stratification factors

5. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of participants who achieved CR as best response and based on Investigator's assessment according to RECIST v 1.1. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
Time Frame: Baseline until disease progression, death or EOT up to data cut-off: 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
percentage of participants | 1 [1 to 6] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Alisertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.283, Weighted Cochran-Mantel-Haenszel test — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.01, 95% CI 2-sided [0.01 to 9999.99] — Logistic regression using CRR as dependent variable, treatment arm as independent variable and disease subtype (sensitive vs resistant/refractory) and presence of brain metastases as stratification factors

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved CR, PR, or SD (when SD was a minimum of 8 weeks in duration). Duration of SD was defined as the time from the date of randomization to the date of first documentation of disease progression for participants who achieved SD as their best overall response. CR was defined as disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker levels. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as ≥ 30% decrease in sum of LD of target lesions in reference to Baseline sum LD. PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline until disease progression, death or EOT up to data cut-off: 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
percentage of participants | 58 [47 to 69] | 46 [35 to 57]
Statistical Analysis 1: Comparison: Alisertib + Paclitaxel vs Placebo + Paclitaxel; Test type: Superiority; p = 0.077, Weighted Cochran-Mantel-Haenszel test — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.32 to 1.08] — Logistic regression using DCR as dependent variable, treatment arm as independent variable and disease subtype (sensitive vs resistant/refractory) and presence of brain metastases as stratification factors

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a PR or better to the date of first documentation of PD for responders. PR was defined as ≥ 30% decrease in sum of longest diameter (LD) of target lesions in reference to Baseline sum LD. PD was defined as ≥20% increase in sum LD in reference to the smallest on-study sum LD, or the appearance of new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first documented response until disease progression until data cut-off 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment. Responders were evaluated for this outcome measure. Responders without documentation of PD were censored at their date of last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 20 | 16
days | 96 [84 to 141] | 85 [58 to 177]

8. Secondary Outcome: Change From Baseline in Symptom (QLQ-LC13 Cough Scale, QLQ-C30 Dyspnea Scale, QLQ-C30 Pain Scale) Score at Cycle 5
Description: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 is 30-item questionnaire with 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (fatigue, nausea, vomiting and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions use 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions use 7-point scale (1=very poor - 7=Excellent). Total Score=0-100 scale; for 5 functional scales and global quality-of-life scale, a higher score=a better level of functioning. For symptoms scale, higher score= higher level of symptoms. EORTC QLQ-LC13 is considered as standard instrument to assess the quality of life (QL) of lung cancer participants. Total Score=0-100. Higher score=increase in level of symptomatology. The change between (QLQ-LC13 Cough Scale, QLQ-C30 Dyspnea Scale, QLQ-C30 Pain Scale) score collected at Cycle 5 relative to baseline.
Time Frame: Baseline up to Cycle 5 (approximately 4.6 months)
Population: The ITT population was defined as all participants who were randomized to study treatment. Here number of participants analyzed are participants evaluated in this outcome measure at the specific timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 20 | 15
score on a scale
  Change at Cycle 5, QLQ-LC-13 Cough Scale | -10.94 (3.07) | 8.07 (6.04)
  Change at Cycle 5, QLQ-C30 Dyspnea Scale | -3.48 (4.25) | -1.09 (2.92)
  Change at Cycle 5, QLQ-C30 Pain Scale | -4.82 (4.86) | -4.88 (5.16)

9. Secondary Outcome: Percentage of Participants Experiencing Symptom Relief
Description: Percentage of participants experiencing symptom relief, including coughing relief, dyspnea relief, and pain relief. Coughing relief is defined as a decrease from baseline ≥ 10 in QLQ-LC13 cough scale/item score. Dyspnea relief is defined as a decrease from baseline ≥ 10 in QLQ-C30 dyspnea scale/item score. Pain relief is defined as a decrease from baseline ≥ 10 in QLQ-C30 pain scale score. EORTC QLQ-C30 is 30-item questionnaire with 5 functional scales, 1 global health status scale, 3 symptom scales, 6 single items. Total Score=0-100 scale; for 5 functional scales and global quality-of-life scale, a higher score=a better level of functioning. For symptoms scale, higher score= higher level of symptoms. EORTC QLQ-LC13 is considered as standard instrument to assess the QL of lung cancer participants. Total Score=0-100. Higher score=increase in level of symptomatology.
Time Frame: Baseline up to Cycle 11, data cut-off: 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment. Participants without coughing/dyspnea/pain relief were censored at their last assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
percentage of participants
  Coughing Relief | 28 [19 to 39] | 24 [15 to 34]
  Dyspnea Relief | 31 [22 to 42] | 16 [9 to 25]
  Pain Relief | 39 [29 to 50] | 36 [26 to 47]

10. Secondary Outcome: Time to Symptom Relief
Description: Time to symptom (coughing/dyspnea/pain) relief was defined as the time from the date of randomization to the date of first detection of coughing/dyspnea/pain relief, respectively.
Time Frame: Baseline up to Cycle 11, data cut-off: 03 January 2016 (approximately 9.8 months)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
months
  Time to Coughing Relief | NA [7.6 to NA] — Median and Upper Limit of Confidence Interval (CI) were not estimable due to low number of participants with events. | NA [NA to NA] — Median, Lower and Upper Limit of CI were not estimable due to low number of participants with events.
  Time to Dyspnea Relief | NA [NA to NA] — Median, Lower and Upper Limit of CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, Lower and Upper Limit of CI were not estimable due to low number of participants with events.
  Time to Pain Relief | 3.0 [1.9 to NA] — Upper Limit of CI was not reached due to low number of participants with events. | 3.7 [1.1 to NA] — Upper limit of CI was not reached due to low number of participants with events.

11. Secondary Outcome: Time to Symptom Progression
Description: Time to coughing/dyspnea/pain progression was defined as time from the date of randomization to date of first detection of progression. Coughing progression was defined as increase from baseline ≥10 in QLQ-LC13 cough scale/item score. Dyspnea progression was defined as increase from baseline ≥10 in QLQ-C30 dyspnea scale/item score. Pain progression was defined as increase from baseline ≥10 in QLQ-C30 pain scale score. EORTC QLQ-C30 is 30-item questionnaire with 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (fatigue, nausea, vomiting and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The QLQ-LC13 is 13-item scale for assessing treatment-specific symptoms in lung cancer. Total Score= 0-100 scale; for 5 functional scales and global quality-of-life scale, higher score=better level of functioning. For symptoms scale, higher score=higher level of symptoms.
Time Frame: Baseline up to Cycle 11, data cut-off: 03 January 2016 (approximately 9.8 months)
Population: The ITT population was defined as all participants who were randomized to study treatment. Participant without coughing/dyspnea/pain progression were censored at their last assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 89 | 89
months
  Time to Coughing Progression | NA [NA to NA] — Median, Lower and Upper Limit of CI were not estimable due to low number of participants with events. | 2.8 [2.2 to 6.3]
  Time to Dyspnea Progression | 3.7 [1.9 to NA] — Upper Limit of CI was not estimable due to low number of participants with events. | 4.6 [1.9 to 6.3]
  Time to Pain Progression | 2.9 [2.1 to NA] — Upper Limit of CI was not estimable due to low number of participants with events. | 2.8 [1.9 to NA] — Upper Limit of CI was not estimable due to low number of participants with events.

12. Secondary Outcome: Observed Plasma Concentration for Alisertib
Time Frame: Day 1 pre-dose and 1, 2-4, 3-6, 10-11 hours post-dose; Day 8, 2 hours post-dose; Day 15, 6-9 hours (hrs) post-dose
Population: Safety population was defined as all participants who received at least 1 dose of any study drug. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Alisertib + Paclitaxel
Number analyzed (Participants) | 87
nM
  Cycle 1, Day 1, Pre-Dose | 0 (0)
  Cycle 1, Day 1, 1 hr Post-Dose: number analyzed (Participants) | 85
  Cycle 1, Day 1, 1 hr Post-Dose | 495.37 (663.456)
  Cycle 1, Day 1, 2-4 hrs Post-Dose: number analyzed (Participants) | 85
  Cycle 1, Day 1, 2-4 hrs Post-Dose | 861.18 (616.951)
  Cycle 1, Day 1, 3-6 hrs Post-Dose: number analyzed (Participants) | 84
  Cycle 1, Day 1, 3-6 hrs Post-Dose | 1048.88 (716.447)
  Cycle 1, Day 1, 10-11 hrs Post-Dose: number analyzed (Participants) | 12
  Cycle 1, Day 1, 10-11 hrs Post-Dose | 539.15 (291.170)
  Cycle 1, Day 8, 2 hrs Post-Dose: number analyzed (Participants) | 76
  Cycle 1, Day 8, 2 hrs Post-Dose | 897.41 (816.387)
  Cycle 1, Day 15, 6-9 hrs Post-Dose (1st Sample): number analyzed (Participants) | 53
  Cycle 1, Day 15, 6-9 hrs Post-Dose (1st Sample) | 1102.93 (612.265)
  Cycle 1, Day 15, 6-9 hrs Post-Dose (2nd Sample): number analyzed (Participants) | 51
  Cycle 1, Day 15, 6-9 hrs Post-Dose (2nd Sample) | 976.92 (572.090)

13. Secondary Outcome: Observed Plasma Concentration for Paclitaxel
Time Frame: Day 1 pre-dose and 1, 2-4, 3-6, 10-11 hours post-dose; Day 8, 2 hours post-dose; Day 15, 6-9 hours post-dose
Population: Due to change in planned analysis, data was only collected and summarized for alisertib not for paclitaxel.
Arm/Group | Alisertib + Paclitaxel
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Biomarker Correlative Studies Including Circulating Tumor Cells and Circulating DNA Assessments
Time Frame: Day 1 cycle 1 in a 28-day cycle
Population: This is an exploratory endpoint.
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: Health Related Quality of Life (HRQOL )
Time Frame: Baseline up to Cycle 11, data cut-off: 03 January 2016 (approximately 9.8 months)
Population: This is an exploratory endpoint.
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after the last dose of study drug (Up to 646 Days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Population included all participants who received at least dose of any study drug.
Arm/Group | Alisertib + Paclitaxel | Placebo + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 12/87 | 11/89
Serious Adverse Events (participants affected / at risk) | 39/87 | 30/89
Other Adverse Events (participants affected / at risk) | 85/87 | 80/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib + Paclitaxel (N=87) | Placebo + Paclitaxel (N=89)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (12) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is related with study drug.
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (3) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is related with study drug.
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is related with study drug.
Septic shock (Infections and infestations) | 1 (1) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is related with study drug.
Pneumonia (Infections and infestations) | 3 (3) | 1 (3) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Pneumocystis jirovecii infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (2) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (7) — Four treatment-emergent deaths occurred during treatment in Placebo + Paclitaxel arm group and are not related with study drug.
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) — Two treatment-emergent deaths occurred during treatment in Alisertib+ Paclitaxel arm group and are not related with study drug.
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) — Two treatment-emergent death occurred during treatment in Alisertib+ Paclitaxel arm group and is not related with study drug.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is not related with study drug.
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 3 (4) | 1 (1) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and two treatment-emergent deaths occurred during treatment in Alisertib + Paclitaxel arm group and are not related with study drug.
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — One treatment-emergent death occurred during treatment in Placebo + Paclitaxel arm group and is not related with study drug.
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (2) | 0 (0) — One treatment-emergent death occurred during treatment in Alisertib + Paclitaxel arm group and is not related with study drug.
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alisertib + Paclitaxel (N=87) | Placebo + Paclitaxel (N=89)
Diarrhoea (Gastrointestinal disorders) | 48 (104) | 18 (32)
Nausea (Gastrointestinal disorders) | 30 (43) | 30 (38)
Vomiting (Gastrointestinal disorders) | 28 (45) | 19 (27)
Stomatitis (Gastrointestinal disorders) | 27 (49) | 6 (7)
Constipation (Gastrointestinal disorders) | 8 (11) | 21 (25)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (7) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 5 (5) | 3 (3)
Fatigue (General disorders) | 38 (52) | 28 (35)
Asthenia (General disorders) | 14 (32) | 11 (16)
Oedema peripheral (General disorders) | 6 (7) | 10 (14)
Pyrexia (General disorders) | 8 (8) | 6 (7)
Non-cardiac chest pain (General disorders) | 4 (5) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 38 (55) | 18 (23)
Neutropenia (Blood and lymphatic system disorders) | 41 (89) | 7 (11)
Leukopenia (Blood and lymphatic system disorders) | 12 (18) | 5 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 29 (36) | 19 (26)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (12) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (23) | 19 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 17 (18)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (10)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 15 (17) | 9 (14)
Headache (Nervous system disorders) | 9 (9) | 6 (7)
Neuropathy peripheral (Nervous system disorders) | 8 (10) | 7 (10)
Paraesthesia (Nervous system disorders) | 4 (5) | 6 (9)
Hypoaesthesia (Nervous system disorders) | 4 (5) | 5 (6)
Somnolence (Nervous system disorders) | 5 (6) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 5 (10)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 6 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (8)
Neutrophil count decreased (Investigations) | 14 (28) | 4 (4)
Weight decreased (Investigations) | 13 (18) | 5 (7)
White blood cell count decreased (Investigations) | 12 (20) | 1 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (15) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (10)
Insomnia (Psychiatric disorders) | 7 (7) | 7 (8)
Confusional state (Psychiatric disorders) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 5 (5) | 11 (13)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.